CLINICAL TRIAL: NCT06545955
Title: A Phase 3, Randomised, Multi-center, Open Label Trial to Evaluate the Safety and Efficacy of Intravesical Nadofaragene Firadenovec Alone or in Combination With Chemotherapy or Immunotherapy in Participants With High-grade Bacillus Calmette-Guerin Therapy (BCG) Unresponsive Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: A Trial to Evaluate Intravesical Nadofaragene Firadenovec Alone or in Combination With Chemotherapy or Immunotherapy in Participants With High-grade BCG Unresponsive Non-muscle Invasive Bladder Cancer
Acronym: ABLE-22
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000434; U1111-1299-0176 (Other: World Health Organization)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Non-muscle Invasive Bladder Cancer With Carcinoma in Situ
MeSH Terms: interventions — Gemcitabine; Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nadofaragene firadenovec (Experimental): Nadofaragene firadenovec (intravesical)
  Interventions: Drug: Nadofaragene Firadenovec
- Nadofaragene firadenovec + gemcitabine & docetaxel (Experimental): Nadofaragene firadenovec (intravesical), and sequential gemcitabine and docetaxel (intravesical)
  Interventions: Drug: Nadofaragene Firadenovec; Drug: Gemcitabine; Drug: Docetaxel
- Nadofaragene firadenovec + pembrolizumab (Experimental): Nadofaragene firadenovec (intravesical), and pembrolizumab (IV infusion)
  Interventions: Drug: Nadofaragene Firadenovec; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nadofaragene Firadenovec — vector-based gene therapy for NMIBC treatment to potentiate durable therapeutic responses by interferon (IFN) alfa-2b (IFN-α2b) amplification. It is a non-replicating recombinant adenovirus serotype 5 vector containing a transgene encoding the human IFN-α2b gene.
  Other Names: ADSTILADRIN
Drug: Gemcitabine — Intravesical Gemcitabine chemotherapy, used in combination with Docetaxel.
  Arms: Nadofaragene firadenovec + gemcitabine & docetaxel
Drug: Docetaxel — Intravesical Docetaxel chemotherapy, used in combination with Gemcitabine.
  Arms: Nadofaragene firadenovec + gemcitabine & docetaxel
Drug: Pembrolizumab — Pembrolizumab is an FDA approved immune checkpoint inhibitor which restores the anti-tumour immune response by blocking the programmed cell death protein 1 (PD-1). Pembrolizumab is administered via intravenous (IV) infusion.
  Arms: Nadofaragene firadenovec + pembrolizumab

SUMMARY:
The pivotal phase 3 trial (rAd-IFN-CS 003) evaluating the efficacy of nadofaragene firadenovec showed that 55 (53.4%) of 103 subjects with CIS ± high-grade Ta/T1 achieved a complete response (CR) at 3 months. In this trial, the safety and efficacy of intravesical instillation of nadofaragene firadenovec alone or in combination with chemotherapy or immunotherapy will be evaluated in participants with NMIBC CIS (± high-grade Ta/T1).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed, as documented, with carcinoma in situ (CIS) ±Ta/T1 high-grade disease.

  * For T1 disease biopsies should contain muscle fibres.
* Unresponsive to ≥2 courses of Bacillus Calmette-Guerin (BCG) therapy within the last 12 months. BCG-unresponsive refers to participants with high-grade non-muscle invasive bladder cancer (NMIBC) who are unlikely to benefit from and who will not be receiving further intravesical BCG. The term "BCG-Unresponsive" includes participants who did not respond to BCG treatment and have a persistent high-grade recurrence within 12 months after BCG was initiated, and those who despite an initial complete response to BCG, relapse with CIS within 12 months of their last intravesical treatment with BCG or relapse with high-grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG. The following criteria define the participants who may be included in the trial:

  * Have received at least 2 courses of BCG within a 12 month period - defined as at least 5 of 6 induction BCG instillations and at least 2 of 3 instillations of maintenance BCG, or at least 2 of 6 instillations of a second induction course, where maintenance BCG is not given.

    o Exception: those who have T1 high-grade disease at 1st evaluation after induction BCG alone (at least 5 of 6 doses) may qualify in the absence of disease progression
  * At the time of tumour recurrence, participants with CIS alone or high-grade Ta/T1 with CIS should be within 12 months of last exposure to BCG
  * No maximum limit to the amount of BCG administered
  * All visible papillary tumours must be resected and those with persistent T1 disease on transurethral resection of bladder tumour (TURBT) should undergo an additional re-TURBT within 14 to 70 days prior to beginning trial treatment. Obvious areas of CIS should also be fulgurated
* Eastern Cooperative Oncology Group (ECOG) status ≤2
* Aged ≥18 years at the time of consent
* Available for the whole duration of the trial
* Life expectancy >2 years, in the opinion of the investigator
* Absence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra. Freedom from upper tract disease (if clinically indicated) as indicated by no evidence of upper tract tumour by either intravenous pyelogram, retrograde pyelogram, computed tomography (CT) scan with or without urogram, or magnetic resonance imaging (MRI) with or without urogram performed within 6 months of enrolment. Absence of locally advanced disease as assessed by CT scan or MRI
* Participants who elect not to undergo cystectomy
* Participants with prostate cancer on active surveillance at low risk for progression are permitted to be included into the trial at the discretion of the investigator
* Females of reproductive potential must have a negative highly sensitive urine or serum pregnancy test upon entry into this trial and be willing to use highly effective contraception during treatment with the investigational medicinal product and for 6 months following the last dose. Otherwise, female participants must be post-menopausal (no menstrual period for a minimum of 12 months, as confirmed by follicle-stimulating hormone levels) or surgically sterile
* Male subjects must use highly effective contraception and a condom during sexual contact regardless of partner's childbearing potential, until 3 months following the last trial drug administration.

Exclusion Criteria:

* Current or previous evidence of muscle-invasive (muscularis propria) or metastatic disease presented at the screening visit. Examples of increased risk of muscle-invasive disease include but are not limited to:

  * Presence of lymphovascular invasion and / or micropapillary, sarcomatoid, plasmacytoid and / or neuroendocrine disease as shown in the histology of the biopsy sample
  * Participants with CIS+T1 disease accompanied by the presence of hydronephrosis secondary to the primary tumour
* Current systemic therapy for bladder cancer other than investigational medicinal products used in randomisation arm
* Current or prior investigational treatment for BCG-unresponsive NMIBC or any other investigational drug (drug used in a clinical trial, i.e drug used in a Ferring sponsored non interventional study does not apply) within 1 month prior to screening
* Current or prior pelvic external beam radiotherapy within 2 years of screening
* Prior treatment with nadofaragene firadenovec at any time
* Prior systemic therapy for bladder cancer at any time
* Prior intravesical chemotherapy for the treatment of BCG-unresponsive NMIBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response | up to 6 months
  Complete response (CR) at any time from first treatment (defined as absence of high-grade (HG) recurrence).

SECONDARY OUTCOMES:
Complete response at month 3 | 3 months
  Complete response 3 months from first treatment
Complete response at month 6 | 6 months
  Complete response 6 months from first treatment
Durability of complete response | Up to 24 months
  Durability of complete response (defined as time from achieved CR to HG recurrence, progression or death due to any cause).
Muscle-invasive progression of disease | up to 36 months
  Muscle-invasive progression of disease (defined as time from first treatment to first evidence of muscle-invasive disease or death)
Cystectomy-free survival | up to 36 months
  Cystectomy-free survival (defined as time from first treatment to either cystectomy or death due to any cause)
Pathological staging | up to 36 months
  Pathological staging (tumor, node, metastasis staging system) in participants at time of cystectomy
Overall survival | up to 36 months
  Overall survival (defined as time from first treatment to death due to any cause)
Evidence of malignant lesions of the upper tract and/or prostatic urethra | up to 24 months
  Evidence of malignant lesions of the upper tract and/or prostatic urethra (defined as time from first treatment to first evidence of malignant lesions).
Adverse events | up to 36 months
  Adverse events collected for nadofaragene firadenovec in combination with chemotherapy (gemcitabine and docetaxel) or immunotherapy (pembrolizumab)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (63):
- United States (33):
  - American Institute of Research, Los Angeles, California
  - USC Kenneth Norris Jr Cancer Hospital, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Genesis Research, LLC - San Diego, San Diego, California
  - Advent Health, Denver, Colorado
  - Colorado Urology - St. Anthony Hospital Campus, Lakewood, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sarasota Memorial Healthcare System, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - Boise VA Medical Center, Boise, Idaho
  - NextStage Clinical Research, Lisle, Illinois
  - Indiana University, Indianapolis, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Atlantic Health, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Great Lakes Physician PC d/b/a Western new York Urology Associates, Cheektowaga, New York
  - Northwell Health -The Arthur Smith Institute for Urology, Lake Success, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine - Penn Urology, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas PLLC (Dallas), Dallas, Texas
  - Houston Methodist Hospital (Houston), Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (2):
  - Prostate Cancer Centre, Calgary, Alberta
  - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
- Czechia (5):
  - Krajska Nemocnice Liberec, Liberec, Liberecký kraj
  - Fakultní Thomayerova Nemocnice, Prague, Prague
  - Fakultni nemocnice v Motole, Prague, Prague
  - Androgeos, spol. s r.o., Prague, Prague
  - Kromerizska Nemocnice A S, Kroměříž, Zlín
- France (8):
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Hospices Civils de Lyon - Edouard Herriot Hosp., Lyon, Auvergne-Rhône-Alpes
  - CHU Toulouse - Hopital Rangueil, Toulouse, Huate-Garonne
  - CHU Nantes - Hotel Dieu, Nantes, Nantes
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire De Nimes (Nîmes), Nîmes, Occitanie
  - Hopital La Pitie Salpetriere, Paris
  - APHP - Hopital Bichat, Paris, Île-de-France Region
- Poland (3):
  - IN-VIVO Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością Medic-R Sp.k., Poznan, Wielkopolska
  - Medical Concierge Centrum Medyczne, Warsaw, Woj. Mazowieckie
- Samsung Medical Center, Seoul, Seoul, South Korea
- Spain (11):
  - Instituto de Investigacion Valdecilla (IDIVAL) / Hospital universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clinic De Barcelona - University of Barcelona, Barcelona, Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario de A Coruna, A Coruña, Galicia
  - Clinica Universidad de Navarra - Madrid, Madrid, Madrid
  - Hospital Universitario 12 De Octubre (Madrid), Madrid, Madrid
  - Universidad Autonoma de Madrid. Hospital Universitario La Paz, Madrid, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Servicio Andaluz de Salud (SAS) - Hospital Universitario Virgen de la Victoria (HUVV), Málaga

IPD SHARING:
Plan to Share IPD: No